CLINICAL TRIAL: NCT05900583
Title: Efficacy Evaluation and Recurrence Monitoring of Neoadjuvant Therapy and Adjuvant Therapy for Esophageal Squamous Cell Carcinoma Based on ctDNA-MRD.
Brief Title: Efficacy Evaluation and Recurrence Monitoring of Therapy for Esophageal Squamous Cell Carcinoma Based on ctDNA-MRD.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Haplox (Unknown)
Responsible Party: Sponsor
Other Study IDs: RICE-MRD
Record Dates: First submitted 2023-05-12; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Minimal Residual Disease; Esophageal Squamous Cell Carcinoma
Keywords: Minimal Residual Disease; Esophageal Squamous Cell Carcinoma; Efficacy Evaluation; Recurrence Monitoring
MeSH Terms: conditions — Neoplasm, Residual; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MRD positive group
- MRD negative group

SUMMARY:
This project is focusing on who have locally advanced esophageal squamous cell carcinoma and have undergone neoadjuvant and adjuvant therapy, followed by surgical resection. The exclusive MRD (Minimal residual disease) probe consists of an exclusive "molecular label" formulated according to the individual genome mutation profile and 21 critical tumor driver genes. By continuously monitoring each patient's ctDNA dynamics, changes in ctDNA concentration or ctDNA-MRD negative/positive results will serve as the primary indicators to assess the efficacy and prognosis of patients with esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
The goal of this project is to recruit 50 patients who have locally advanced esophageal squamous cell carcinoma and have undergone neoadjuvant and adjuvant therapy, followed by surgical resection. Initially, tumor tissues from all patients will undergo a more comprehensive NGS sequencing process (WESPlus) than whole-exome sequencing. This will provide a complete genomic mutation profile for each patient. Subsequently, a specific algorithm will be used to accurately select 20 mutation sites as the patient's unique "molecular label." Additionally, 21 critical driver genes related to tumors will be combined, leading to the creation of an exclusive MRD probe. This will enable ultra-high-depth capture sequencing of ctDNA samples from patients at 100,000x. By continuously monitoring each patient's ctDNA dynamics, changes in ctDNA concentration or ctDNA-MRD negative/positive results will serve as the primary indicators to assess the efficacy and prognosis of patients with esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 80 years old;
* Patients diagnosed with locally advanced esophageal squamous cell carcinoma by imaging or pathological examination: cT2-4N1-3M0, cT3-4N0M0 II-IVA (including IVB stage with supraclavicular and abdominal lymph node metastasis);
* Receive neoadjuvant therapy;
* Must be able to obtain the patient's clinical information and clear pathological diagnosis results;
* Able to cooperate with long-term follow-up, regular review, and blood sample collection;
* Patients agree to participate in the tracking and follow-up of the group and provide follow-up information;
* Must obtain the informed consent of the patient or their legal representative, and the patient has the ability to cooperate to complete the requirements of the study.

Exclusion Criteria:

* Patients with other cancers or severe illnesses that result in shorter survival than the trial follow-up period;
* Received other treatments (such as radiotherapy, etc.) before receiving neoadjuvant therapy;
* Have contraindications to chemotherapy;
* Patients who received blood transfusions within three months prior to enrollment;
* HIV-positive patients or those with other immune system deficiency diseases;
* Pregnant patients;
* Alcohol or drug abusers;
* Other situations that the researchers believe may affect the experimental results or are unethical.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced esophageal squamous cell carcinoma by imaging or pathological examination: cT2-4N1-3M0, cT3-4N0M0 II-IVA (including IVB stage with supraclavicular and abdominal lymph node metastasis);.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | immediately after surgery
  No residual tumor is the esophagus or dissected lymph nodes.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | 2 years
  The time from date of diagnosis to the time of recurrence or death.
Overall survival (OS) | 2 years
  The time from date of diagnosis to the time of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No